CLINICAL TRIAL: NCT01787292
Title: Effects of Exercise Intervention on Aging-related Motor Decline (AGING)
Brief Title: Effects of Exercise Intervention on Aging-related Motor Decline
Acronym: EIAMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: E0956-W; 2012-060697 (Other Grant/Funding Number: Veterans Affairs)
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Aging; Exercise
Keywords: Exercise; Magnetic Resonance Imaging; Transcranial Magnetic Stimulation; Aging
MeSH Terms: conditions — Motor Activity | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: A. Light stretching and balance exercises under supervised trainer. 3 times per week for 20-45 minutes. HR will be targeted to be under 50% of age-related maximum.
  B. Interval aerobic cycling under supervised trainer. 3 times per week for 20-45 minutes. HR will be targeted between 50-85% of age-related maximum.
  C. 6 month self-monitored training phase during which time participants will exercise using a take home bike ergometer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stretching Exercise Intervention (Experimental): A. Light stretching and balance exercises under supervised trainer. 3 times per week for 20-45 minutes. HR will be targeted to be under 50% of age-related maximum.
  Interventions: Behavioral: Stretching Exercise Intervention
- Aerobic Exercise Intervention (Experimental): B. Interval aerobic cycling under supervised trainer. 3 times per week for 20-45 minutes. HR will be targeted between 50-85% of age-related maximum.
  Interventions: Behavioral: Aerobic Exercise Intervention
- Self Monitoring Intervention (Experimental): C. 6 month self-monitored training phase during which time participants will exercise using a take home bike ergometer.
  Interventions: Behavioral: Self Monitoring

INTERVENTIONS:
Behavioral: Stretching Exercise Intervention — A. Light stretching and balance exercises under supervised trainer. 3 times per week for 20-45 minutes. HR will be targeted to be under 50% of age-related maximum.
  Arms: Stretching Exercise Intervention
Behavioral: Aerobic Exercise Intervention — Supervised weekly exercise. 3 bouts of 45 minutes weekly on a cycle ergometer. HR will be kept at 75% of age-related maximum.
  Arms: Aerobic Exercise Intervention
Behavioral: Self Monitoring — 6 month self-monitored training phase during which time participants will exercise according to prescribed regimen (cycling)
  Arms: Self Monitoring Intervention

SUMMARY:
The purpose of this research study is to test whether differing levels of physical fitness affects patterns of motor dexterity and brain activity that have been shown to differ due to aging. Testing will take place at the Atlanta VA Medical Center and at Emory University.

Participants will be healthy adults within the target age range of 60-85 for the study. The study will require multiple visits over 15 months. There will be about 64 people volunteering for this study.

DETAILED DESCRIPTION:
The U.S. Census reports over 14 million U.S. Veterans (>63%) are beyond mid-life (>55 years). Declines in upper extremity motor performance respective of strength and dexterity are well documented within this age cohort). Recent cross-sectional research has discovered that aging related motor deficits may be influenced by a loss of interhemispheric inhibition (IHI) between primary motor cortices. However, this loss may not be an inevitable consequence of aging. Work from previous VA OAA Predoctoral and CDA-1 awards have shown that aerobic fitness may serve to mitigate losses in interhemispheric inhibition assessed by both functional magnetic resonance imaging (fMRI) and transcranial magnetic stimulation (TMS). That is, individuals who are aerobically fit show higher levels of IHI and improved dexterity and reaction times.

In light of new evidence from the investigators' lab's recent cross-sectional studies, physical activity over the long term (at least 2-5 years) may serve to alter levels of IHI and improve motor performance in the upper extremity. Aerobic exercise may provide a mechanism (reduced loss of interhemispheric inhibition) that could serve to improve motor function, but the neural mechanism responsible for such effects remains unclear. Previous investigations of interhemispheric communication and exercise have been limited by nature of inquiry, as cross-sectional research cannot measure changes over time in participants. As such, it is currently unknown how exercise may directly affect levels of interhemispheric communication and motor performance.

Behavioral interventions (motor strength and coordination) have been shown to be effective in improving upper extremity motor performance in older adults, however the duration of these gains appear to be short-lived. After as little as a few weeks of detraining, motor strength and coordination in the upper extremity rapidly begins to return to pre-intervention levels. Evidence from exercise interventions assessing gait and locomotion have shown that exercise programs over a longer term (>6 months) are associated with improved proprioception, fewer falls and better balance. However, the comparison of outcomes of upper extremity function in elderly adults respective of exercise duration remains largely unexplored. In addition to comparing the effects of short-term exercise (3 months) versus behavioral training (3 months) on upper extremity function, the current proposal will evaluate if a longer-term (6 months) exercise program can maintain or enhance upper extremity function and associated levels of interhemispheric inhibition.

The current study proposes the next logical step in my line of research and directly investigates the effects of exercise in an intervention with sedentary older Veterans (50-80 years), a group most likely to exhibit aging-related motor deficits. The investigators propose to enroll 40 Veterans into an upper extremity dexterity improvement program involving behavioral and exercise components. The behavioral intervention is a muscle coordination training previously shown to improve unimanual motor performance in older adults. The exercise intervention is a supervised group cycling regimen. The figure below shows the study design. Interhemispheric communication will be assessed with fMRI, and TMS.

ELIGIBILITY:
Inclusion Criteria:

* Living persons between 60 and 85 years of age

Exclusion Criteria:

* unmanaged diabetes
* participants completing vigorous exercise per week
* participants whose profession requires vigorous physical labor
* contraindication to magnetic resonance imaging

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith M. McGregor, PhD MS BA, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McGregor KM, Crosson B, Mammino K, Omar J, Garcia PS, Nocera JR. Influences of 12-Week Physical Activity Interventions on TMS Measures of Cortical Network Inhibition and Upper Extremity Motor Performance in Older Adults-A Feasibility Study. Front Aging Neurosci. 2018 Jan 4;9:422. doi: 10.3389/fnagi.2017.00422. eCollection 2017. PMID 29354049
- [Result] Nocera J, Crosson B, Mammino K, McGregor KM. Changes in Cortical Activation Patterns in Language Areas following an Aerobic Exercise Intervention in Older Adults. Neural Plast. 2017;2017:6340302. doi: 10.1155/2017/6340302. Epub 2017 Mar 6. PMID 28367334
- [Result] McGregor KM, Crosson B, Krishnamurthy LC, Krishnamurthy V, Hortman K, Gopinath K, Mammino KM, Omar J, Nocera JR. Effects of a 12-Week Aerobic Spin Intervention on Resting State Networks in Previously Sedentary Older Adults. Front Psychol. 2018 Nov 27;9:2376. doi: 10.3389/fpsyg.2018.02376. eCollection 2018. PMID 30542314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community-dwelling individuals were recruited for participation using approved flyer and advertising materials. All participants gave voluntary written consent prior to participation. After consenting, participants were randomly assigned to one of two 12-week exercise interventions involving a followed by cross-over to the other intervention.
Groups:
- Experimental: Aerobic Exercise, Then Balance Training: Participants completed a 12-week interval aerobic cycling under supervised trainers three times per week for 20-45 minutes per session. After two to four week washout period, participants entered a second 12-week intervention involving light stretching and balance exercise under a supervised trainer three times per week for 20-45 minutes per session.
- Experimental: Balance Training, Then Aerobic Exercise: Participants completed a 12-week light stretching and balance exercise program under a supervised trainer three times per week for 20-45 minutes per session.Participants completed an interval aerobic cycling under supervised trainer three times per week for 20-45 minutes per session. After two to four week washout period, participants completed a 12-week interval aerobic cycling under supervised trainers three times per week for 20-45 minutes per session.
Period: Crossover Exercise Interventions
Arm/Group | Experimental: Aerobic Exercise, Then Balance Training | Experimental: Balance Training, Then Aerobic Exercise
Started | 17 (Participants in this group performed aerobic training prior to cross-over to balance training.) | 16 (Participants in this group performed balance training prior to cross-over to aerobic training.)
Completed | 15 (Participants completed the 12-week in-house program and cross-over into the balance program.) | 14 (These participants completed the 12-week in-house program and cross-over into the balance program.)
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Home Based Exercise Program
Arm/Group | Experimental: Aerobic Exercise, Then Balance Training | Experimental: Balance Training, Then Aerobic Exercise
Started | 15 | 14
Completed | 12 | 13
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Exercise Interventions for Crossover Design: This study was a cross-over design with two groups to which participants were randomized. Group one received a 12-week Aerobic exercise intervention and then crossed over into a balance exercise intervention. Group two received the balance intervention for 12 weeks and then crossed over into the aerobic exercise intervention. All completing participants then engaged in a home based exercise program during which they were instructed to exercise thrice weekly over 24 weeks.
Arm/Group | Exercise Interventions for Crossover Design
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.05 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Cardiovascular Efficiency [Mean (Standard Deviation); unit: ml/kg(min)] | 25.25 (9.74)
Ipsilateral Silent Period [Mean (Standard Deviation); unit: milliseconds] | 22.39 (4.73)
FMRI of Right Motor Cortex [Mean (Standard Deviation); unit: area under curve] | 1.85 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Estimate Cardiovascular Efficiency After Aerobic Exercise
Description: Estimate of Volume of oxygen consumption (VO2peak) using YMCA protocol for cardiovascular assessment.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Estimated VO2 peak values in ml/kg(min)
Measure: Mean (Standard Deviation); unit: ml/kg(min)
Groups:
- Experimental: Aerobic First: Aerobic Exercise: Interval based spin exercise under a supervised trainer three times per week for 20-45 minutes per session.
Arm/Group | Experimental: Aerobic First
Number analyzed (Participants) | 15
ml/kg(min)
  Baseline | 24.01 (9.29)
  12-Week post | 31.2 (8.6)
  24-week post-cross | 32.3 (6.8)
Statistical Analysis 1: Comparison: Experimental: Aerobic First; Test type: Superiority; p = .001, ANCOVA — To account for sequence carryover, we employed analysis of covariance inclusive of sequence by period covariates against treatment effects; Least square means were adjusted for carryover from the crossover design and between subjects effects were analyzed using Kenward-Roger df estimation

2. Primary Outcome: Estimate of Cardiovascular Efficiency After Balance Training
Description: Estimated VO2peak using YMCA cycle test completed over nine to twelve minutes.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Sedentary older adults who engaged in less than 45 minutes of regular exercise per week
Measure: Mean (Standard Deviation); unit: ml/kg(min)
Groups:
- Balance Training: Effects of Balance/Stretching training after 12-week intervention
Arm/Group | Balance Training
Number analyzed (Participants) | 14
ml/kg(min)
  Pre | 22.83 (7.35)
  12-Weeks | 24.72 (9.36)
  24-week post-cross | 23.58 (8.25)
Statistical Analysis 1: Comparison: Balance Training; To account for sequence carryover, we employed analysis of covariance inclusive of sequence by period covariates against treatment effects; Test type: Superiority; p = .8, ANCOVA

3. Primary Outcome: Silent Period Duration After Exercise Cycling Program
Description: Duration of ipsilateral silent period from Transcranial magnetic stimulation measured in milliseconds
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Exercise - Cycling: Short Term exercise - supervised: Supervised weekly exercise. 3 bouts of 45 minutes weekly on a cycle ergometer. HR will be kept at 75% of age-related maximum.
Arm/Group | Exercise - Cycling
Number analyzed (Participants) | 15
milliseconds
  Baseline | 22 (7.8)
  12-Week post | 26.2 (7.5)
  24-week post-cross | 27.5 (7.4)
Statistical Analysis 1: Comparison: Exercise - Cycling; Test type: Superiority; p = .05, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Silent Period Duration for Balance Group
Description: Ipsilateral silent period duration as assessed by TMS
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Sedentary older adults engaging in less than 45 minutes of total activity per week
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Balance Training
Number analyzed (Participants) | 14
milliseconds
  Pre | 23 (8.9)
  12-Weeks | 21.2 (5.1)
  24-week post-cross | 26.2 (8.1)
Statistical Analysis 1: Comparison: Balance Training; Test type: Superiority; p = .05, ANCOVA — [p-value comment as in outcome 1, analysis 1]; A Kenward-Rogers adjustment for degrees of freedom was made to account for carryover effects

5. Primary Outcome: fMRI Interhemispheric Inhibition Improvement After Aerobic Exercise
Description: Participants who exercise will evidence larger increases in interhemispheric inhibition as assessed by functional magnetic resonance measured by a z-normalized area under curve of right primary motor cortex. The area under the curve is an estimate of the fMRI hemodynamic response impulse response function. A higher number of AUC indicates less interhemispheric inhibition. In contrast, a lower number in this analysis indicates higher interhemispheric inhibition.
Time Frame: Baseline to 24 Weeks with cross-over
Population: Analysis of area under curve of right primary motor cortical area
Measure: Mean (Standard Deviation); unit: Z-transformed impulse response function
Groups:
- Aerobic First Then Balance Cross-over: Aerobic cycling first then cross-over to balance group
Arm/Group | Aerobic First Then Balance Cross-over
Number analyzed (Participants) | 15
Z-transformed impulse response function
  Pre | 1.5 (1.2)
  12 week intervention | .58 (.98)
  24 week post-crossover | .58 (.98)
Statistical Analysis 1: Comparison: Aerobic First Then Balance Cross-over; Test type: Superiority; p = .01, t-test, 2 sided

6. Primary Outcome: fMRI Interhemispheric Inhibition Improvement After Balance Training
Description: Area under the curve of fMRI measures of right motor cortex BOLD profile will remain similar to pre measurements. The BOLD profile is the z-normalized area under the curve value of the fMRI impulse response function. A higher number indicates less interhemispheric inhibition.
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: Z-transformed impulse response function
Arm/Group | Balance Training
Number analyzed (Participants) | 14
Z-transformed impulse response function
  Pre | 1.49 (.88)
  12-Weeks | .62 (.52)
  24-week post-cross | .62 (.52)
Statistical Analysis 1: Comparison: Balance Training; Test type: Superiority; p = .01, t-test, 2 sided

7. Primary Outcome: Comparison of Cardiovascular Efficiency for Aerobic Exercise First Group After Home-based Intervention
Description: Comparison of home based aerobic exercise intervention to assessments made after completion of crossover intervention in Participants receiving aerobic condition first. VO2peak estimation completed using the YMCA protocol investigating overall volume of oxygen consumption as a function of heart rate during work loads. Estimated VO2 peak values are in ml/kg(min).
Time Frame: 24 and 48 weeks
Measure: Mean (Standard Deviation); unit: ml/kg(min)
Arm/Group | Exercise Interventions for Crossover Design
Number analyzed (Participants) | 12
ml/kg(min)
  Within one week of completing 24 week intervention | 25.25 (12.25)
  Within one week of completing 48 Week Intervention | 21.2 (9.88)
Statistical Analysis 1: Comparison: Exercise Interventions for Crossover Design; Test type: Superiority; p = .01, t-test, 2 sided

8. Primary Outcome: Comparison of Cardiovascular Efficiency for Balance Exercise First Group After Home-based Intervention
Description: VO2peak estimation completed using the YMCA protocol investigating overall volume of oxygen consumption as a function of heart rate during work loads.
Time Frame: 24 and 48 weeks
Population: Participants completed both exercise interventions but completed Balance training prior to engaging in aerobic exercise training.
Measure: Mean (Standard Deviation); unit: ml/kg(min)
Groups:
- Balance Training: Effects of Balance/Stretching training after study completion
Arm/Group | Balance Training
Number analyzed (Participants) | 12
ml/kg(min)
  Within one week of completing 24 week intervention | 25.5 (12.8)
  Within one week of completing 48 Week Intervention | 20.8 (12.2)
Statistical Analysis 1: Comparison: Balance Training; Test type: Superiority; p = .5, t-test, 2 sided

9. Primary Outcome: Comparison of Silent Period Duration After Aerobic Exercise
Description: Comparison of silent period duration at 24 weeks compared to baseline
Time Frame: Baseline, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Aerobic Exercise: Participants in this group first received a 12-week Aerobic exercise intervention and then crossed over into a balance exercise intervention.
Arm/Group | Aerobic Exercise
Number analyzed (Participants) | 15
milliseconds
  Pre | 20.58 (7.5)
  12-Weeks | 26.2 (7.5)
  24-week post-cross | 27.5 (7.4)
Statistical Analysis 1: Comparison: Aerobic Exercise; Test type: Superiority; p = .6, t-test, 2 sided; A Kenward-Rogers adjustment for df was made to account for carryover effects

10. Primary Outcome: Comparison of Silent Period Duration After Balance Exercise
Description: Comparison of Home based training effects on TMS measures of silent period duration as compared to facility based exercise programs.
Time Frame: 24 and 48 weeks
Population: Participants completing balance training then crossing over into aerobic exercise were then tested for effects of facility based treatments against home exercise.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Balance Training
Number analyzed (Participants) | 12
milliseconds
  Within one week of completing 24 week intervention | 26.54 (8.4)
  Within one week of completing 48 Week Intervention | 21.6 (9.3)
Statistical Analysis 1: Comparison: Balance Training; Test type: Superiority; p = .4, t-test, 2 sided

11. Secondary Outcome: Target Heart Rate Zone for Balance First Participants
Description: Heart rate in aerobic target zone is measured in percentage of time in at least 50% of participants heart rate reserve.
Time Frame: 24 and 48 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Balance Training
Number analyzed (Participants) | 14
percentage of time
  Within one week of completing 24 week intervention | 58.4 (34.6)
  Within one week of completing 48 Week Intervention | 88.5 (14.7)
Statistical Analysis 1: Comparison: Balance Training; Test type: Superiority; p = .05, t-test, 2 sided

12. Secondary Outcome: Target Heart Rate Zone After Aerobic Exercise First
Description: Targeted Heart Rate Zone among participants compared among short term exercise groups
Time Frame: 24 and 48 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Exercise - Cycling
Number analyzed (Participants) | 15
percentage of time
  Within one week of completing 24 week intervention | 93.7 (10.1)
  Within one week of completing 48 Week Intervention | 70.6 (22.5)
Statistical Analysis 1: Comparison: Exercise - Cycling; Test type: Superiority; p = .25, t-test, 2 sided

13. Secondary Outcome: Heart Rate Workload After Home Based Intervention
Description: Measured heart rate after home based intervention
  Technical implementation at the facility level prevented acquisition of these metrics until late in the project.
Time Frame: 24 and 48 weeks
Population: Participants completing home based interventions compared to facility based interventions - measured in time in aerobic zone.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Exercise Interventions for Crossover Design
Number analyzed (Participants) | 7
percentage of time
  Within one week of completing 24 week intervention | 78 (18)
  Within one week of completing 48 Week Intervention | 48 (30)
Statistical Analysis 1: Comparison: Exercise Interventions for Crossover Design; Test type: Superiority; p = .01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 60 month. Participants were assessed at baseline, after 12-weeks, after 24 weeks and after 48 weeks. Measurements at 12 weeks represent first intervention. Measurements at 24 weeks represent measure after cross-over into alternate intervention. All participants then went through a home-based exercise program, which is the 48 week assessment. Note: Participants may have withdrawn from the study prior to completing the home-based exercise program.
Groups:
- Experimental Intervention: Aerobic Exercise First: Participants completed a 12-week interval aerobic cycling under supervised trainers three times per week for 20-45 minutes per session. After two to four week washout period, participants entered a second 12-week intervention involving light stretching and balance exercise under a supervised trainer three times per week for 20-45 minutes per session.
  Participants later crossed over into the Balance condition and were assessed at 24 weeks.
  After this time, participants completed a 24 week home based aerobic exercise program. This intervention was common to both groups and therefore are collapsed within this Arm.
- Experimental Intervention: Balance Exercise First: Participants completed a 12-week light stretching and balance exercise program under a supervised trainer three times per week for 20-45 minutes per session.Participants completed an interval aerobic cycling under supervised trainer three times per week for 20-45 minutes per session. After two to four week washout period, participants completed a 12-week interval aerobic cycling under supervised trainers three times per week for 20-45 minutes per session.
  Participants later crossed over into the Aerobic Exercise condition and were assessed at 24 weeks.
  After this time, participants completed a 24 week home based aerobic exercise program. This intervention was common to both groups and therefore are collapsed within this Arm.
Arm/Group | Experimental Intervention: Aerobic Exercise First | Experimental Intervention: Balance Exercise First
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

LIMITATIONS AND CAVEATS:
Local procurement difficulties limited remote tracking of participants in 6-month home exercise arm of program. This caused lower-than-expected adherence and negatively affected long-term outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT01787292/Prot_SAP_000.pdf